CLINICAL TRIAL: NCT01790230
Title: LifeSeal™ Preliminary Study in Subjects Undergoing Low Anterior Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeBond Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLP-LS-0105
Record Dates: First submitted 2013-01-31; First posted 2013-02-13 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- Standard of Care (No Intervention): Standard of Care Arm - subjects treated by routine manner
- LifeSeal™ Kit (Experimental): LifeSeal™ Kit Arm - subjects treated with the LifeSeal™ Kit device + Standard of Care treatment
  Interventions: Device: LifeSeal™ Kit

INTERVENTIONS:
Device: LifeSeal™ Kit — Application of LifeSeal™ Kit for staple line reinforcement during open GI surgeries in Low Anterior Resection
  Arms: LifeSeal™ Kit

SUMMARY:
A preliminary Study in Subjects Undergoing Low Anterior Resection

ELIGIBILITY:
Inclusion Criteria:

1. Subject, or authorized representative, signed a written Informed Consent
2. Subject is at least 18 years of age
3. Subject is scheduled for elective open resection
4. Stapled anastomosis created within 10cm of the anal verge
5. Subject is willing to comply with the follow-up requirements of the study

Exclusion Criteria:

1. Subject has a history of hypersensitivity to porcine derived gelatin or collagen
2. Subject has unacceptable baseline hematological results
3. Subject on chronic preoperative treatment with steroids and anticoagulants
4. Subject with elevated liver function tests
5. Subject with abnormal kidney function
6. Subject with a BMI higher than 35
7. Subject participating in any other study for either drug or device which can influence collection of valid data under this study
8. Subject with a history of MI, CVA or ASA status IV or a life expectancy of less than 1 year
9. Anastomosis was performed differently from what was defined
10. Subject received intraoperative sealant, glue or any buttressing material for the study related anastomosis, other than the LifeSeal™
11. Subject has intraoperative bleeding in excess of 500cc
12. Subject has peritoneal carcinomatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Assessment of subject's safety by incidence of related Adverse Events | Approx. 1 month

SECONDARY OUTCOMES:
Assessment of the device's application technique | Intra-operative
  Surgeon will complete a questionnaire regarding the device use and ease of application

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden